CLINICAL TRIAL: NCT05864872
Title: What is the Best Approach for Blocking Intercostobrachial and Medial Brachial Cutaneous Nerves in the Upper Arm Surgery? Ultrasound as an Alternative to Blind Infiltration
Brief Title: the Best Approach for Blocking Intercostobrachial and Medial Brachial Cutaneous Nerves in the Upper Arm Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olfa kaabachi, MD (Other)
Responsible Party: Sponsor-Investigator, Olfa kaabachi, MD, MD, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: olfakaabachi
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2024-02

CONDITIONS: Pain
Keywords: brachial plexus block; ultrasound; infiltration
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): after blockage of the principal four nerves of the brachial plexus, the needle was redirected, and between 1 and 2 mL of bupivacaine was injected around each visible nerve branch (Intercostobrachial and Medial Brachial Cutaneous ); if the nerve branches were not visible, 5 mL of the local anesthetic was injected (or less volume if the nerves appeared during the injection), in the subcutaneous area located above the brachial fascia, with a posterior direction, toward the latissimus dorsi muscle.
  Interventions: Procedure: axillary brachial plexus block
- conventional group (Active Comparator): after blockage of the principal four nerves of the brachial plexus, 3 to 6 mL of bupivacaine (at the discretion of the anesthesiologist) was infiltrated blindly subcutaneously at the same level of the axilla in the anteroposterior direction prior to complete needle withdrawal
  Interventions: Procedure: axillary brachial plexus block

INTERVENTIONS:
Procedure: axillary brachial plexus block — conventional group, 3 to 6 mL of bupivacaine was infiltrated blindly subcutaneously at the same level of the axilla in the anteroposterior direction prior ultrasound group:1 and 2 mL of bupivacaine was injected around each visible nerve branch (Intercostobrachial and Medial Brachial Cutaneous ); if the nerve branches were not visible, 5 mL of the local anesthetic was injected in the subcutaneous area located above the brachial fascia, with a posterior direction, toward the latissimus dorsi muscle.
  Other Names: conventional group; ultrasound group

SUMMARY:
Brachial plexus block (BPB) alone, whether performed at the axilla or more proximally, does not provide sufficient anesthesia for the skin of the medial upper arm and elbow, because thoracic roots contribute to the innervation of these areas.

For surgery of the upper arm, the brachial plexus block needs to be completed by the Medial Brachial Cutaneous nerve (MBCN) and the Intercostobrachial nerve (ICBN) nerve blocks.

The ICBN is not part of the brachial plexus; it usually originates from the lateral branch of the second intercostals nerve (T2). The MBCN and the ICBN are often interconnected. In the axilla, they are separated from the brachial plexus by the brachial fascia. Therefore, when an axillary brachial plexus block (ABPB) is performed, the local anesthetic solution may be prevented from spreading toward the MBCN and ICBN.

These nerves are classically anesthetized by raising a subcutaneous wheel of local anesthetic spanning the entire width of the medial aspect of the arm at the level of the axilla, usually from anteriorly to posteriorly. The failure rate of this blind infiltration procedure has never been quantified in the literature. Traditional teaching suggests that the ICBN should be blocked to prevent tourniquet pain. Lanz et al (1) showed that BPB, whether performed to the axilla or more proximally, rarely extend to the ICBN (10% of cases). However, recent literature shows differences in opinion on the role of an ICBN/MBCN blocks in preventing tourniquet pain. Ultrasound guided ABPB is sufficient to provide anaesthesia for tourniquet even during prolonged ischemia. However, to ensure prevention of tourniquet discomfort a multiple injection technique that include musculocutaneous blockade should be preferred (2). The overall incidence of tourniquet pain in the setting of an effectively dense supraclavicular brachial plexus block for surgical anesthesia was low, even without the addition of an ICBN block. This tourniquet pain can be easily managed with small increases in systemic analgesics (3). However, in Magazzeni Ph et al (4) study, ultrasound-Guided Block of ICBN and MBCN was associated to a better sensory block and a less painful tourniquet compared to conventional block.

The optimal access for an ultrasound guided block of the MBCN and the ICBN nerves is not yet known.

DETAILED DESCRIPTION:
* Routine monitoring was applied, and intravenous access secured for each patient.
* Sedation with 2 mg of midazolam was administrated
* 2L of O2 were administrated through nasal cannula
* Physical separation between the patient and the anesthesiologist was established before the block procedure
* Ultrasound images were acquired with SonoSite(Turbo M), and a linear ultrasound probe (6-13 MHz) was used.
* Nerve blocks were performed with 100mm 22-gauge needles (Braun), in an awake patient through ideally a single skin puncture.
* In both groups, the median, radial, ulnar, musculocutaneous, and medial antebrachial cutaneous nerves were blocked with a total of 30 mL of a mixiture of 0.5 %bupivacaine + 1% lilocaine
* Intraoperatively, if the tourniquet was painful, fentanyl and additional midazolam dose were administered.

Patients are allocated to one of the two groups:

Group C In patients allocated to the conventional group, 3 to 6 mL of bupivacaine (at the discretion of the anesthesiologist) was infiltrated blindly subcutaneously at the same level of the axilla in the anteroposterior direction prior to complete needle withdrawal.

Group U In patients allocated to the USG group, the needle was redirected, and between 1 and 2 mL of bupivacaine was injected around each visible nerve branch (MBCN and ICBN); if the nerve branches were not visible, 5 mL of the local anesthetic was injected (or less volume if the nerves appeared during the injection), in the subcutaneous area located above the brachial fascia, with a posterior direction, toward the latissimus dorsi muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patient belonged to (ASA) physical status 1 2 3, aged more than 18 years old and scheduled for surgery of the upper limb (hand, forearm, elbow, and anteromedial and posteromedial arm).

Exclusion Criteria:

* Patients refusal, any allergy to the study drugs, local infection at any of the puncture sites, any coagulation disorder, or any neurological or psychological problem which may have affected proper subjective interpretation of the results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
tourniquet pain | during surgery
  The proportion of patients pain free when inflating tourniquet.

SECONDARY OUTCOMES:
sensitive block | 5, 10, 15 and 20 minutes after performing the block
  The proportion of patients who had no sensation in all 4 regions innervated by both Intercostobrachial and Medial Brachial Cutaneous Nerves
rescue sedetion | during surgery
  Proportion of patient with rescue sedation/analgesia because of uncomfortable tourniquet
durationof ultrasound image | during ultrasound procedure
  time to ultrasound visualisation of both Intercostobrachial and Medial Brachial Cutaneous Nerves
Quality of ultrasound images | during ultrasound procedure
  visualization of the 2 nerves

CONTACTS AND LOCATIONS:
Locations (1):
- KAABACHI, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No